CLINICAL TRIAL: NCT02420236
Title: Effects of Resistance Training on Pain, Function and Work Ability in Patients With Moderate to Severe Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other); Kommunal Landspensjonskasse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1157-B
Record Dates: First submitted 2015-03-18; First posted 2015-04-17 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Low Back Pain
Keywords: Exercise therapy; Resistance training; Multidisciplinary treatment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity resistance training (Experimental): Full body, progressive strength training with Theraband® Elastic bands. Three times per week for 12 weeks - 3 weeks with supervised sessions at the clinic, and 9 weeks of home training. Three guided sessions will be offered during the home training period.
  Interventions: Behavioral: High-intensity resistance training; Behavioral: Multidisciplinary rehabilitation program
- General physical activity (Active Comparator): 12 weeks of general physical activity - 3 weeks with supervised sessions at the clinic, and 9 weeks of individually adjusted home training. This include circle-training, low-intensity resistance exercises, endurance exercises, ball playing, body awareness, stretching, and relaxation techniques, and similar activities. Neither moderate nor high-intensity resistance exercise is included for participants in this group.Three guided sessions will be offered during the home training period.
  Interventions: Behavioral: General physical activity; Behavioral: Multidisciplinary rehabilitation program

INTERVENTIONS:
Behavioral: High-intensity resistance training
  Arms: High-intensity resistance training
Behavioral: General physical activity
  Arms: General physical activity
Behavioral: Multidisciplinary rehabilitation program

SUMMARY:
The purpose of this study is to investigate if high-intensity resistance training can induce additional beneficial effects, for patients with moderate to severe long term pain in the low back, when added to a multidisciplinary treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the multidisciplinary clinic for treatment of pain in low back
* Long term (≥ 3months) or recurrent (≥ 2 periods of ≥ 4 weeks the past year) non-specific low back pain
* Pain intensity ≥ 4 on numerical rating scale (0-10)

Exclusion Criteria:

* Severe somatic condition (unstable injury, malignity, infectious disease, active rheumatic disease, severe osteoporosis)
* Psychiatric condition/disease that severely impairs group functioning
* Insufficient comprehension of Norwegian language to participate in group sessions and fill out questionnaires
* Awaiting surgery of back
* Alcohol or drug abuse
* Ongoing compensation case or applying for disability benefits due to pain in the back
* Engaged in high-intensity resistance training on a regular basis the last 6 months

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Low back-related disability as assessed by the oswestry disability index | 12 weeks
  Oswestry disability index

SECONDARY OUTCOMES:
Pain assessed by the Numerical Pain Rating Scale | 3 and 12 weeks + 6 and 12 months
Fear avoidance beliefs assessed by Fear Avoidance Beliefs Questionnaire | 3 and 12 weeks + 6 and 12 months
Patients' perceived effect of the treatment assessed by the Patient specific functioning scale | 3 and 12 weeks + 6 and 12 months
Anxiety and depression assessed by Hopkins symptom checklist | 3 and 12 weeks + 6 and 12 months
Quality of life assessed by EQ-5D-5L | 3 and 12 weeks + 6 and 12 months
Work ability assessed by Work ability index | 3 and 12 weeks + 6 and 12 months
Use of analgesics assessed by a questionnaire from the HUNT study | 3 and 12 weeks + 6 and 12 months
Physical activity level assessed by a questionnaire from the HUNT study | 3 and 12 weeks + 6 and 12 months
Strength in the low back during maximal isometric contractions of the back extensors | 3 and 12 weeks + 6 and 12 months
Grip strength using a handheld dynamometer | 3 and 12 weeks + 6 and 12 months
Patients' perceived effect of the treatment assessed by the Global rating of change scale | 3 and 12 weeks + 6 and 12 months
Low back-related disability as assessed by the oswestry disability index | 3 weeks + 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marius S Fimland, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs University Hospital - Department of Physical Medicine and Rehabilitation, Trondheim, Norway

REFERENCES:
- [Background] Iversen VM, Vasseljen O, Mork PJ, Berthelsen IR, Borke JB, Berheussen GF, Tveter AT, Salvesen O, Fimland MS. Resistance training in addition to multidisciplinary rehabilitation for patients with chronic pain in the low back: Study protocol. Contemp Clin Trials Commun. 2017 Apr 12;6:115-121. doi: 10.1016/j.conctc.2017.04.001. eCollection 2017 Jun. PMID 29740641
- [Result] Iversen VM, Vasseljen O, Mork PJ, Gismervik S, Bertheussen GF, Salvesen O, Fimland MS. Resistance band training or general exercise in multidisciplinary rehabilitation of low back pain? A randomized trial. Scand J Med Sci Sports. 2018 Sep;28(9):2074-2083. doi: 10.1111/sms.13091. Epub 2018 Apr 24. PMID 29603805